CLINICAL TRIAL: NCT06389513
Title: Phase IV Clinical Study of the Safety of Menhycia® in 3-Month-Old Infants
Brief Title: Clinical Study of the Safety of Menhycia® in 3-Month-Old Infants
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CTP-MCVF-005
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Epidemic Meningitis
Keywords: Vaccine; ACYW135; CRM197; Safety; 3 months of age
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197) (MCV4) (Experimental): Intramuscular injection, 0.5ml
  Interventions: Biological: MCV4

INTERVENTIONS:
Biological: MCV4 — 4 doses of vaccine on Day 0, Day30, Day 60 and Month 12

SUMMARY:
This study is an open, multicenter Phase IV clinical study to evaluate the safety of vaccination with Menhycia®. The study plan is to enroll approximately 3,000 infants at 3 months of age who have not been vaccinated with any epidemic encephalitis vaccine, and to administer a total of 3 doses of Menhycia®, with a minimum of 1 month between doses, and a booster dose of 1 dose of immunization is allowed at 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Infants 3 months of age who had not received any epidemic encephalitis vaccine at the time of screening
* The legal guardian or delegate has given informed consent, has voluntarily signed an informed consent form, and is able to comply with the requirements of the clinical study protocol

Exclusion Criteria:

First dose exclusion criteria

* Fever before vaccination, axillary temperature >37.0°C
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* History of epilepsy, convulsions or seizures or history or family history of psychiatric disorders
* Acute infections or active chronic diseases, severe infectious or allergic skin diseases
* Known allergy to a component of the vaccine, especially to diphtheria toxoid, or to previous administration of the product
* Other circumstances that, in the judgment of the investigator, make participation in this clinical study inappropriate

Subsequent dose exclusion criteria

* Severe allergic reactions after a previous dose of vaccine
* Those with serious adverse reactions causally related to the previous dose of vaccination
* Other circumstances that, in the judgment of the investigator, make participation in this clinical study inappropriate

Ages: 3 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3011 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of localized adverse reactions in subjects | Within 7 days after each dose of vaccination
Incidence of systemic adverse reactions in subjects | Within 7 days after each dose of vaccination

SECONDARY OUTCOMES:
Incidence of adverse reactions in subjects | Within 30 days after each dose of vaccination
Incidence of adverse events in subjects | Within 30 days after each dose of vaccination
Incidence of severe adverse events | Through study completion, an average of 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Luhe District Center for Disease Control and Prevention Center for Disease Control and Prevention, Nanjing, China